CLINICAL TRIAL: NCT00438126
Title: Family-Centered Diabetes Project - Sharing Wisdom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DK47096 (completed)
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Prediabetes; Metabolic Syndrome; Overweight; Obesity
Keywords: diabetes; Prevention; American Indian
MeSH Terms: conditions — Prediabetic State; Metabolic Syndrome; Overweight; Obesity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: A lifestyle educational program

SUMMARY:
This is a randomized trial of an educational intervention to reduce the risk of diabetes among urban American Indian women

DETAILED DESCRIPTION:
Two hundred American Indian women aged 18 to 40 years were recruited from a large Southwest city to participate in a type 2 diabetes prevention intervention. Half of the women were randomized to participated in the educational intervention and half were assigned to a delayed intervention. Measures were obtained at baseline, 6-months,12-months and 18-months.

ELIGIBILITY:
Inclusion Criteria:

* American Indian women
* Aged 18-40 years
* Living in Albuquerque area
* Not having diabetes

Exclusion Criteria:

* Pregnancy
* Planning to become pregnant within 2 years
* Diagnosed with diabetes fasting blood glucose > 126 planning to move out of town in next 2 years

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200
Dates: Start 2002-01; Study Completion 2006-05

PRIMARY OUTCOMES:
decreased dietary fat intake
increased vegetable consumption
increased self-reported leisure physical activity

SECONDARY OUTCOMES:
fasting glucose
HOMA
serum free insulin
Body Mass Index
waist circumference
decreased dietary intake of total sugar
decreased time watching television
resting blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Herman, MD, MPH, Principal Investigator — Univeristy of New Mexico
Locations (1):
- University of New Mexico School of Medicine, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Willging CE, Helitzer D, Thompson, J 'Sharing Wisdom': Lessons learned during the development of a diabetes prevention intervention for urban American Indian women Evaluation and Program Planning 29 (2006) 130-140
- [Background] Helitzer D, Peterson AB, Thompson J, Fluder S. Development of a planning and evaluation methodology for assessing the contribution of theory to a diabetes prevention lifestyle intervention. Health Promot Pract. 2008 Oct;9(4):404-14. doi: 10.1177/1524839906289076. Epub 2006 Jul 21. PMID 16861598
- [Derived] Thompson JL, Allen P, Helitzer DL, Qualls C, Whyte AN, Wolfe VK, Herman CJ. Reducing diabetes risk in American Indian women. Am J Prev Med. 2008 Mar;34(3):192-201. doi: 10.1016/j.amepre.2007.11.014. PMID 18312806